CLINICAL TRIAL: NCT04930419
Title: Comparative Evaluation of the McGrath Videolaryngoscope and the Direct Laryngoscopy for Tracheal Intubation in the Prehospital Setting
Acronym: AMAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K170405J
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Indication of Orotracheal Intubation; Cardio Respiratory Arrest; Respiratory Failure; Neurological Failure
MeSH Terms: conditions — Heart Arrest; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscopy group (Other)
  Interventions: Device: Videolaryngoscopy group
- Direct laryngoscopy group (Other)
  Interventions: Device: Direct laryngoscopy group

INTERVENTIONS:
Device: Videolaryngoscopy group — Tracheal intubation will be performed using Videolaryngoscope in first intention and will be performed using standard pre-hospital intubation procedures : preoxygenation before intubation, maintenance of oxygenation throughout procedure, standard sedation technique (using rapid sequence intubation (RSI)), correct position confirmation using a capnogram and conditioning (hemodynamic monitoring, respirator settings, securing). If the first attempt at intubation is unsuccessful, further management will be left to the discretion of the clinician according to the procedures and algorithm of usual standard care
  Arms: Videolaryngoscopy group
Device: Direct laryngoscopy group — Tracheal intubation will be performed using Direct laryngoscopy with Macintosh blades in first intention. and will be performed using standard pre-hospital intubation procedures : preoxygenation before intubation, maintenance of oxygenation throughout procedure, standard sedation technique (using rapid sequence intubation (RSI)), correct position confirmation using a capnogram and conditioning (hemodynamic monitoring, respirator settings, securing). If the first attempt at intubation is unsuccessful, further management will be left to the discretion of the clinician according to the procedures and algorithm of usual standard care
  Arms: Direct laryngoscopy group

SUMMARY:
In the prehospital setting, the risk of difficult intubation and life-threatening complications is increased under particular conditions due to the environment or the frequent instability of patients.

To limit this risk procedures and devices to ease and secure tracheal intubation must be developped and integrated.

As the prevalence of complications increase with the number of attempts of intubation, one strategy is to facilitate the intubation technic itself.

Direct laryngoscopy with Macintosh blades is the standard device commonly used in first place for tracheal intubation.

Other devices are available and used, mostly for difficult intubation, included videolaryngoscopy. This device has been used and studied for years now. Allowing a better view and glottic visualisation, videolaryngoscopy could increase the first-pass success rate.

Among all videolaryngoscopes, the McGrath videolaryngoscope is the most similar device to the standard Macintosh laryngoscope. It is light, compact, with a screen directly linked to the handle, easy to use and offering excellent view. Its usability and efficacy make it a device of choice for the prehospital setting and worth further clinical trials to define its place in the airway strategy.

Hypothesis: In the prehospital setting, the use of McGrath videolaryngoscope as the primary device for tracheal intubation could facilitate tracheal intubation and decrease the number of attempts of intubation and complications.

The objective of our study is to determine if the use of McGrath videolaryngoscope increase the rate of successful first-pass intubation in the prehospital setting compared to direct view Macintosh laryngoscopy.

The primary outcome is the rate of successful intubation at the first attempt. One attempt is defined as an advancement of the tube towards the glottis during a laryngoscopy ; every new try even during the same laryngoscopy is considered as a new attempt.

Successful intubation is confirmed by the visualisation of 6 waves of EtCO2.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18
* Indication of orotracheal intubation
* Operators trained to the use of the McGrath

Exclusion Criteria:

* Pregnancy
* No insurance
* Major patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of successful intubation at the first attempt | up to 10 minutes post inclusion
  One attempt is defined as an advancement of the tube towards the glottis during a laryngoscopy ; every new try even during the same laryngoscopy is considered as a new attempt.Successful intubation is confirmed by the visualisation of 6 waves of EtCO2.

SECONDARY OUTCOMES:
Number of attempts needed for successful intubation | up to 10 minutes post inclusion
Time to intubate | up to 10 minutes post inclusion
  Time to intubate will be defined by the time between the insertion of the device in the mouth and the visualisation of the first waves of EtCO2
Reason of failure of the first-pass success | up to 10 minutes post inclusion
  Reasons of failure will be defined as following :
  * Bad glottic visualization
  * Difficult progression of the tube towards the glottis despite a good visualisation
  * Presence of secretions
  * Presence of foreign body
  * Presence of fogging on the McGrath
  * Device failure
  * Other
Proportion of decision of switch in case of failure | up to 10 minutes post inclusion
Proportion of difficult intubations | up to 10 minutes post inclusion
  Difficult intubation will be evaluated by the intubation difficulty score (score IDS or difficulty of intubation under laryngoscopy score ). It goes from 0 to infinity. zero indicating an easy intubation and infinity being an impossible intubation
Glottic view | up to 10 minutes post inclusion
  Glottic view will be evaluated with Cormack and Lehane grade and POGO score. POGO score goes from 0 (Visualization of the language base) to 100% (total visualization of the glottis). Cormack and Lehane grade goes from I to IV. A higher Cormack and Lehane grade is worth : I indicate total visualization of the glottis and IV indicate Visualization of the language base
Proportion of cases who need for tools to optimize | up to 10 minutes post inclusion
Proportion of cases needed crossovers to other rescue techniques | up to 10 minutes post inclusion
Number of complications per and post-intubation | up to 10 minutes post inclusion
Type of complications per and post-intubation | up to 10 minutes post inclusion
Number of deaths | up to 10 minutes post inclusion

IPD SHARING:
Plan to Share IPD: Undecided